CLINICAL TRIAL: NCT04145388
Title: Systems-Level Capture of Family History Data to Assess Risk of Cancer
Brief Title: Family History Study on Cancer Risk
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1407426
Record Dates: First submitted 2019-09-30; First posted 2019-10-30 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Lynch Syndrome; Colorectal Cancer; Breast Cancer; Ovarian Cancer; Family Characteristics; Genetic Predisposition
Keywords: cancer; family characteristics; genetic predisposition; primary care
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Colorectal Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Genetic Predisposition to Disease; Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Comparator 1 (Other): Participants will have their cancer risk assessed via usual care. Usual Care is defined as provider capture of family history during a clinical encounter and its entry into the electronic health record (EHR). Participants will take the a patient reported outcomes (PRO) survey once to assess participants experience, perspectives and thoughts on cancer, cancer risk, and cancer risk assessments.
  Interventions: Other: Usual care
- Comparator 2 (Experimental): Participants will have their cancer risk assessed using a short, standardized web-based questionnaire that will populate validated cancer risk models (such as Breast Cancer Risk Assessment Tool/Gail model 2, PREMM and/or MMRpro) which will take 5-10 minutes to complete. Following the cancer risk assessment, participants will be asked to take a PRO survey. PRO surveys will also be administered at the time of the cancer risk assessment and then 6 and 12 months following.
  Interventions: Other: online cancer risk assessment
- Comparator 3 (Experimental): Participants will have their cancer risk assessed using a more detailed, full version of the family history survey than the one comparator 2 participants take. This version is a full pedigree assessment, which entails family health history for all 1st, 2nd, and 3rd-degree relatives. Time needed for completion is 15-25 minutes, depending on family size and cancer risk. Participants will also be asked to take the PRO survey following the full cancer risk assessment and also at 6 and 12 months.
  Interventions: Other: online cancer risk assessment

INTERVENTIONS:
Other: online cancer risk assessment — Electronic surveys to collect family cancer history information.
  Arms: Comparator 2; Comparator 3
Other: Usual care — Family cancer history captured by provider during a clinical encounter
  Arms: Comparator 1

SUMMARY:
This study aims to identify the optimal method to recognize, risk stratify, and provide follow-up care for individuals at risk of hereditary cancer. The study team will conduct a Hybrid Type II comparative effectiveness-implementation trial, with a mixed methods component and process/formative evaluations for stakeholder engagement. The study team will evaluate three methods for identifying and risk-stratifying individuals at risk of hereditary cancer and providing post-risk stratification longitudinal care.

DETAILED DESCRIPTION:
The study team proposes a randomized, Hybrid Type II comparative effectiveness-implementation trial, with a mixed methods component and process/formative evaluations for stakeholder engagement. The study team will evaluate three methods for identifying and risk-stratifying individuals at risk of hereditary cancer and providing post-risk stratification longitudinal care.

Hypothesis: The study hypothesis is that Comparator 3 will identify more people at high risk of hereditary cancers and result in more screening behaviors, greater resource use, increased distress, higher perceived risk of cancer and higher satisfaction.

Long term objective: At study end, the study will show: 1) each comparator's strengths and weaknesses, 2) patient preferences, clinical outcomes, and compliance with each step from history collection to screening test completion, 3) the resources needed for each strategy, and 4) the contextual factors that impact their sustainability, dissemination and implementation. Study findings have high potential for generalizability because: 1) The multidisciplinary stakeholder team will help to minimize barriers to dissemination and implementation of the investigator's findings in other research settings; 2) Study results are independent of study setting; 3) The tested methods of family history assessment can occur remotely via paper or electronic interfaces; 4) The care coordination method has successful precedent in other disciplines and can be delivered remotely; 5) A process and formative evaluation with a diverse stakeholder team will inform sustainability, dissemination, and implementation, and result in an implementation guide; 6) The results will be relevant for both family history-based and direct-genetic testing strategies for population screening for hereditary cancer; 7) The results will inform population screening for any disease with hereditary risk.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with ≥2 years of prior membership, ≥1 clinical visit in prior two years, and a listed email are eligible
* Patients must also have received healthcare services during the past 2 years at Kaiser Permanente Northern California (KPNC) sampling sites

Exclusion Criteria:

* Patients outside the targeted geographic area
* Patients who cannot speak or read English (given some survey instruments are validated only in English)
* Kaiser Permanente Northern California members in the no-contact database for research studies

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18623 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients identified at high risk of cancer | 0 to 12 months
  Number of patients identified at high risk of cancer (cancer syndromes)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Corley, MD, PhD, Principal Investigator — Division of Research, Kaiser Permanente Northern California
Locations (1):
- Division of Research, Kaiser Permanente Northern California, Oakland, California, United States